CLINICAL TRIAL: NCT07366541
Title: Predicting High-Flow Nasal Cannula Failure Using an Electrical Impedance Tomography-Derived Index: A Multicenter Study
Status: Active, not recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20250232
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure; Oxygen Therapy Failure; High-flow Nasal Cannula (HFNC) Therapy; Electrical Impedance Tomography (EIT)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HFNC Oxygen Therapy
  Interventions: Device: Electrical impedance tomography(PulmoVista 500, Dräger Medical)

INTERVENTIONS:
Device: Electrical impedance tomography(PulmoVista 500, Dräger Medical) — Outcome Parameters: FI, ROX index, respiratory rate, SpO₂

SUMMARY:
High-Flow Nasal Cannula (HFNC) therapy is widely used to treat acute respiratory failure. However, predicting therapy failure remains challenging as conventional indices rely on intermittent measurements and cannot provide continuous, objective monitoring. Electrical Impedance Tomography (EIT) enables non-invasive, real-time assessment of regional lung ventilation. This study evaluated whether an EIT-derived Flow Index (FI) could predict HFNC therapy failure within 48 hours.

DETAILED DESCRIPTION:
Design: Single-center, prospective observational study. Setting: Ruijin Hospital, Shanghai, China. Population: Adult patients with acute respiratory failure receiving HFNC between December 2023 and March 2024. Intervention: EIT monitoring during spontaneous breathing while on HFNC. FI was calculated from EIT-derived regional ventilation signals using a curve-fitting formula quantifying inspiratory flow-time waveform concavity.

Endpoints: Primary - HFNC failure (escalation to mechanical ventilation or persistent hypoxemia within 48 h). ROC analysis compared FI with ROX index, respiratory rate, and SpO₂. Logistic regression models assessed predictive value and odds ratios.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Acute respiratory failure requiring HFNC
* Stable hemodynamics
* FiO₂ ≤0.6

Exclusion Criteria:

* Neuromuscular disease affecting spontaneous breathing
* Pregnancy
* Contraindications to EIT
* Poor EIT signal quality

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with acute respiratory failure receiving HFNC
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
HFNC Failure Rate | Within 48 hours of HFNC initiation

SECONDARY OUTCOMES:
ROC comparison of FI, ROX index, and conventional parameters | Within 48 hours
Odds ratio and confidence interval for FI predicting HFNC failure | Within 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hongping Qu, Study Chair — Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of Critical Care Medicine，Ruijin Hospital，Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided